CLINICAL TRIAL: NCT00886041
Title: Role of Laparoscopy in Unexplained Infertility
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: professor ahmed m badawy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: mansoura university
Record Dates: First submitted 2009-04-21; First posted 2009-04-22 (Estimated); Last update posted 2009-04-22 (Estimated); Status verified 2009-04

CONDITIONS: Infertility
Keywords: laparoscopy; unexplained infertility
MeSH Terms: conditions — Infertility | interventions — Laparoscopy; Ovulation Induction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- laparoscopy group (Other): laparoscopy
  Interventions: Procedure: laparoscopy
- ovarian stimulation group (Active Comparator): ovarian stimulation and timed intercourse for 3 cycles followed by ovarian stimulation and intrauterine insemination for another 3 cycles
  Interventions: Other: ovarian stimulation

INTERVENTIONS:
Procedure: laparoscopy — subjected to laparoscopy
  Arms: laparoscopy group
Other: ovarian stimulation — ovarian stimulation and timed intercourse for 3 cycles followed by ovarian stimulation and intrauterine insemination for another 3 cycles
  Arms: ovarian stimulation group

SUMMARY:
In this randomized controlled trial the investigators were looking for the best policy for management of women with unexplained infertility after normal hysterosalpingogram (HSG). The investigators test the hypothesis that postponing or even bypassing laparoscopy does not affect the outcome of management of women with apparently unexplained infertility.

ELIGIBILITY:
Inclusion Criteria:

* failure of conception for at least one year
* no pathology demonstrated after the standard infertility work-up including semen analysis, mid-luteal serum progesterone for confirming ovulation and hysterosalpingography for documenting tubal patency
* diagnosed as having unexplained infertility

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 512 (Actual)
Dates: Start 2003-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The outcome measure was the occurrence of clinical pregnancy and miscarriage. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: ahmed m badawy, MD PhD, Principal Investigator — Mansoura University
Locations (1):
- Mansoura University Hospitals, Al Mansurah, Dakahalia, Egypt